CLINICAL TRIAL: NCT02307227
Title: Antitumor Immune Responses in Breast Cancer Patients Treated With Neoadjuvant Chemotherapy: a Phase II Study With Trastuzumab and Concomitant Weekly Paclitaxel in Patients With HER2+ Tumors or Epirubicin + Taxotere in HER2- Tumors.
Brief Title: Phase II Study With Trastuzumab + Paclitaxel in Locally Advanced HER2+ Tumors or Epirubicin + Taxotere in HER2- Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRO-18-2006
Record Dates: First submitted 2014-11-26; First posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Paclitaxel; Epirubicin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Locally advanced HER2+ breast cancer pts (Experimental): HER2 positive (defined as 3+ at Herceptest or FISH/CISH positive):
  treatment with Trastuzumab 4mg/kg first time, then 2 mg/kg weekly with concomitant paclitaxel 80 mg/mq weekly (one cycle corresponding to 4 weeks) for 12 weeks (3 cycles). Clinical and instrumental evaluation, in responding patients continue for additional 12 weeks (total 6 cycles), then surgical excision
  Interventions: Drug: Trastuzumab; Drug: Paclitaxel
- Locally advanced HER2- breast cancer pts (Experimental): HER2 negative:
  treatment with Epirubicin 90 mg/mq and docetaxel 75 mg/mq every 3 weeks for 4 cycles. Clinical and instrumental evaluation, in responding patients continue for additional 12 weeks (total 8 cycles), then surgical excision.
  Interventions: Drug: Epirubicin; Drug: Docetaxel

INTERVENTIONS:
Drug: Trastuzumab
  Arms: Locally advanced HER2+ breast cancer pts
Drug: Paclitaxel
  Arms: Locally advanced HER2+ breast cancer pts
Drug: Epirubicin
  Arms: Locally advanced HER2- breast cancer pts
Drug: Docetaxel
  Arms: Locally advanced HER2- breast cancer pts

SUMMARY:
Prospective, monoinstitutional, phase II study. Patients with HER 2 positive locally advanced breast cancer will be treated with 3 initial cycles (12 weeks) of trastuzumab plus paclitaxel and then if responding further 12 weeks and then with surgical resection, patients with HER2 negative breast carcinoma will be treated with 4 cycles (12 weeks) of epirubicin and taxotere. If responding 4 more cycles (12 weeks). Patients progressing will be treated depending on physician's and patient's preference

DETAILED DESCRIPTION:
Primary Objective: to determine the pathological complete response (pCR) and correlation with immune response.

Secondary Objectives:

* to determine the progression free survival (PFS) and overall survival (OS);
* to evaluate the safety of the treatment with particular attention to cardiac safety.

Inclusion Criteria:

* Histologically proven breast carcinoma evaluated for HER 2 status and immune status
* Locally advanced carcinoma (UICC stage II-III)
* Age < 70 years
* measurable lesions
* ECOG Performance Status 0-2
* Life expectancy > 3 months
* Adequate bone marrow and hepatic functions
* Creatinine Clearance > 40 ml/min
* Written informed consent
* Patients must be accessible for treatment and follow up

Exclusion criteria:

* Prior chemotherapy or hormonal treatments
* Brain metastases.
* Past or current history of neoplasm other than curatively treated.
* Concurrent treatment with other experimental drugs.
* Left Ventricular Ejection Fraction (LVEF) <50 %
* History of significant neurological or psychiatric disorders.

Treatment HER2 positive (defined as 3+ at Herceptest or FISH/CISH positive) Herceptin 4mg/kg first time, then 2 mg/kg weekly with concomitant paclitaxel 80 mg/mq weekly (one cycle corresponding to 4 weeks) for 12 weeks (3 cycles). Clinical and instrumental evaluation, in responding patients continue for additional 12 weeks (total 6 cycles), then surgical excision

HER2 negative:

Epirubicin 90 mg/mq and docetaxel 75 mg/mq every 3 weeks for 4 cycles. Clinical and instrumental evaluation, in responding patients continue for additional 12 weeks (total 8 cycles), then surgical excision.

Main Parameters of Activity:

* Complete Remission (CR): complete disappearance of all previously detectable disease for a period of at least 28 days, and no new lesions.
* Partial Remission (PR): more than 30% reduction in the longest diameter of target lesions, and no new lesions.
* Stable Disease (SD): less than 30% reduction and less than 20% increase in the longest diameter of target lesions and no new lesions.
* Progressive Disease (PD): an increase in size of more than 20% of at least one lesion of previously documented disease. Or the appearance of disease at any site.
* Progression Free Survival (PFS) will be measured from the first day of the treatment until the first observation of disease progression or death due to any cause or the last date the patient was known to be progression free and alive.
* Overall Survival (OS) will be computed as the time between the first day of treatment and the date of death or the last date the patient was known to be alive.

Main Parameters of Safety:

* Adverse events, laboratory parameters.
* All toxicity will be graded using the NCI common toxicity criteria (Appendix II). Cardiac events (CHF) will be graded according to NYHA

Study procedure:

* At Baseline:
* Complete medical history, ECOG PS, physical examination (including a neurological examination, height, weight,),
* ECG
* Left ventricular ejection fraction evaluation (LVEF, evaluated by echocardiography).
* Blood chemistry (fasting blood sugar, transaminases, serum alkaline phosphatase, total bilirubin, total protein, albumin, creatinine, PT, fìbrinogen)
* Complete blood count and differential
* Calculated Creatinine Clearance/24 h
* Chest X- ray
* Abdomen computer tomography (CT) or ultrasound
* Bone scan and X-ray (if appropriate)
* Written informed consent.
* During Treatment - Every Cycle:
* Blood chemistry
* Complete blood count and differential
* Toxicity evaluation
* Physical examination
* During Treatment - Every 12 weeks (3-4 cycles):
* Breast ultrasound
* Surgical and medical evaluation
* Left ventricular ejection fraction evaluation (LVEF) evaluated by echocardiography
* ECOG PS
* Before surgery:
* Mammography, Ultrasound and Magnetic resonance
* Long term Follow up - Every 3 months for the first 2 years, every 6 months years 3-5 then yearly
* Survival

Statistical Considerations:

The aim of this phase II clinical trial is to detect 20% improvement in the pCR (i.e., from 25% to 54%). Simon's methods will be used to calculate sample size. Accrual of 46 patients has been planned considering a 80% of power to detect a 20% difference (two-sided type I error =0.05). The Chi-square test and Fisher's exact test will be used for qualitative parameters.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven breast carcinoma evaluated for HER 2 status and immune status
* Locally advanced carcinoma (UICC stage II-III)
* Age < 70 years
* measurable lesions
* ECOG Performance Status 0-2
* Life expectancy > 3 months
* Adequate bone marrow and hepatic functions
* Creatinine Clearance > 40 ml/min
* Written informed consent
* Patients must be accessible for treatment and follow up.

Exclusion Criteria:

* Prior chemotherapy or hormonal treatments
* Brain metastases.
* Past or current history of neoplasm other than curatively treated.
* Concurrent treatment with other experimental drugs.
* Left Ventricular Ejection Fraction (LVEF) <50 %
* History of significant neurological or psychiatric disorders.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-04; Primary Completion 2009-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | 60 months
  pCR was defined as no evidence of microscopic residual invasive cancer, both in breast and ipsilateral axillary lymph nodes, or residual carcinoma in situ in the absence of invasive breast cancer

SECONDARY OUTCOMES:
Progression free survival | 60 months
  From the first day of treatment to progression or death due to any cause or last contact patient was to be known progression free or alive
Overall survival | 60 months
  Time between the date of first day of treatment and the date of death from any cause or the last date the patient was known to be alive.
Cardiac safety | 60 months
  Number of patients with adverse cardiac events. The intensity of clinical adverse events will be graded according to the NCI Common Toxicity Criteria grading system in the toxicity categories that have recommended gradings
Host immune response | 60 months
  Multiple parameters were investigated: T-cell responses against 13 immunogenic HLA-A*0201-restricted nonamer (9-mer) peptides; Immune cells subsets (CD3+ T cells, CD19+ B cells, CD3-CD16+CD56+ NK cells, CD3+CD4+ T cells, CD3+CD8+ T cells, CD3+CD4+CD25+CD127-/lowFoxP3+ Treg cells, CD3+CD4+IL17+ Th17 cells. Among CD3+CD4+ and CD3+CD8+ T cells, CCR7+CD45RA+ naïve T cells , CCR7+CD45RA- Central Memory T cells, CCR7-CD45RA- Effector Memory T cells , CCR7-CD45RA+ Terminally Differentiated T cells, trastuzumab-dependent ADCC in the HER-2+ arm. Measure of immunologic parameters: changes from baseline recorded at 12 and 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Dolcetti, MD, Principal Investigator — Centro di Riferimento Oncologico - Aviano
Locations (1):
- Centro di Riferimento Oncologico, Aviano, Pordenone, Italy

REFERENCES:
- [Background] Muraro E, Martorelli D, Turchet E, Miolo G, Scalone S, Comaro E, Talamini R, Mastorci K, Lombardi D, Perin T, Carbone A, Veronesi A, Crivellari D, Dolcetti R. A different immunologic profile characterizes patients with HER-2-overexpressing and HER-2-negative locally advanced breast cancer: implications for immune-based therapies. Breast Cancer Res. 2011;13(6):R117. doi: 10.1186/bcr3060. PMID 22112244
- [Derived] Muraro E, De Zorzi M, Miolo G, Lombardi D, Scalone S, Spazzapan S, Massarut S, Perin T, Dolcetti R, Steffan A, De Re V. KIR-HLA Functional Repertoire Influences Trastuzumab Efficiency in Patients With HER2-Positive Breast Cancer. Front Immunol. 2022 Jan 12;12:791958. doi: 10.3389/fimmu.2021.791958. eCollection 2021. PMID 35095867
- [Derived] Muraro E, Comaro E, Talamini R, Turchet E, Miolo G, Scalone S, Militello L, Lombardi D, Spazzapan S, Perin T, Massarut S, Crivellari D, Dolcetti R, Martorelli D. Improved Natural Killer cell activity and retained anti-tumor CD8(+) T cell responses contribute to the induction of a pathological complete response in HER2-positive breast cancer patients undergoing neoadjuvant chemotherapy. J Transl Med. 2015 Jun 27;13:204. doi: 10.1186/s12967-015-0567-0. PMID 26116238
- [Derived] Miolo G, Muraro E, Martorelli D, Lombardi D, Scalone S, Spazzapan S, Massarut S, Perin T, Viel E, Comaro E, Talamini R, Bidoli E, Turchet E, Crivellari D, Dolcetti R. Anthracycline-free neoadjuvant therapy induces pathological complete responses by exploiting immune proficiency in HER2+ breast cancer patients. BMC Cancer. 2014 Dec 15;14:954. doi: 10.1186/1471-2407-14-954. PMID 25512030